CLINICAL TRIAL: NCT02292810
Title: Acute Effects of Inspiratory Muscle Exercise on Glucose Level and Glucose Variability in Patients With Type 2 Diabetes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 14-0194
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory muscle exercise (Experimental): Patients will exercise the inspiratory muscle using a load of 60% of maximum inspiratory mouth pressure (MIP 60%).
  Interventions: Device: Inspiratory muscle exercise
- Inspiratory muscle exercise placebo (Placebo Comparator): Patients will exercise the inspiratory muscle using a load of 2% of maximum inspiratory mouth pressure (MIP 2%).
  Interventions: Device: Inspiratory muscle exercise placebo

INTERVENTIONS:
Device: Inspiratory muscle exercise — For inspiratory muscle exercise patients will breathe with a high load of 60% of MIP using a respiratory frequency of 15 breaths min and a prolonged duty cycle (TI/TTOT =0.7) until task failure. The blood flow, conductance and resistance arterial will be measured in the calf using plethysmography device. Arterial blood pressure and heart rate will be monitored continuously at the finger on a beat-by-beat basis by biopac equipment and the glucose levels will be captured by continuous glucose monitoring system.
  Arms: Inspiratory muscle exercise
Device: Inspiratory muscle exercise placebo — For inspiratory muscle exercise patients will breathe with a very low load of 2% of MIP using a respiratory frequency of 15 breaths min and a prolonged duty cycle (TI/TTOT =0.7) for 10 minute. The blood flow, conductance and resistance arterial will be measured in the calf using plethysmography device. Arterial blood pressure and heart rate will be monitored continuously at the finger on a beat-by-beat basis by biopac equipment and the glucose levels will be captured by using the continuous glucose monitoring system.
  Arms: Inspiratory muscle exercise placebo

SUMMARY:
Type 2 diabetes is associated with respiratory muscle weakness and autonomic neuropathy. The exercise of inspiratory muscles has been investigating in various clinical situations and may cause similar benefits as the conventional exercises. The assessment of glucose variability has been used as an alternative tool to evaluate the others mechanisms than the absolute values of glucose levels, special during the exercise. However, the effect of inspiratory muscle exercise on glucose levels and glucose variability is not clear yet. The aim of the proposed research is to evaluate the acute effects of inspiratory muscle exercise using a high load of 60% of MIP on glucose levels and glucose variability in patients with type 2 diabetes.

DETAILED DESCRIPTION:
High-intensity exercise of inspiratory muscle was able to reduce glucose levels in previous studies, but the mechanisms underlying this reduction remain largely unknown. The present study will investigate this phenomenon, and whether confirmed, the inspiratory muscle loading would be a new approach for lowering glucose levels and glucose variability in type 2 diabetes.

The subjects with type 2 diabetes will be recruited from the ambulatory of the Hospital de Clinicas de Porto Alegre. The patients will be randomized to inspiratory muscle exercise with a high intensity load (MIP 60%) or to exercise with a load placebo (MIP 2%), on two different days. The subjects will come in the laboratory for three days consecutively during 2 weeks. On the first day will be placed the CGMS device. On the second day will be the controlled ventilation protocol with subsequently inspiratory muscle exercise, using 2% or 60% of MIP as randomized a priori. On the third day the CGMS will be removed. Individuals who are using beta-blockers will be advised to withdraw the medication 24 hours before the protocols. During all protocols will be recorded the continuous blood pressure to assess heart rate and blood pressure variabilities, both time and frequency domains will be analyzed. Also, the calf blood flow, inspiratory pressure, end-tidal carbon dioxide and oxygen saturation will be taking.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* HbA1c from 7,5 to 10%;

Exclusion Criteria:

* Subjects taking insulin;
* Pregnant women;
* Subjects taking betablocker only
* Documented arrythmia
* Documented fibrillation
* GFR<30
* Documented pulmonary disease or asthma,
* Current smoking;
* Varicose vein problems;
* Musculoskeletal disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Glucose level | 1 day (A session of inspiratory muscle exercise)
  The glucose level will be assessed by continuous glucose monitoring (CGMS) before and after exercise.

SECONDARY OUTCOMES:
Glucose variability | 3 days
  The variability of the glucose will be assessed by continuous glucose monitoring (CGMS) 24 hours before exercise, during the protocol and 24 hours after exercise.
Autonomic control | 1 day (A session of inspiratory muscle exercise)
  The autonomic control will be evaluated in the time domain and frequency through the Biopac.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Schaan, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre

REFERENCES:
- [Derived] Schein A, Correa A, Casali KR, Schaan BD. Are glucose levels, glucose variability and autonomic control influenced by inspiratory muscle exercise in patients with type 2 diabetes? Study protocol for a randomized controlled trial. Trials. 2016 Jan 20;17:38. doi: 10.1186/s13063-016-1156-0. PMID 26790405